CLINICAL TRIAL: NCT07333287
Title: A Multicenter Single-arm Prospective Clinical Study on First-line Treatment of Pancreatic Cancer Liver Metastases With Arterial Infusion Chemotherapy and Embolization Combined With Dual Immune Checkpoint Inhibitors.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Dan Sha, Chief Physician, Shandong Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO.2025-1074
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer Liver Metastases; Immunotherapy-naive
MeSH Terms: interventions — Methods; Immunotherapy; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Interventional Combined Targeted Therapy、 Immunotherapy + Targeted Therapy、Immunotherapy + Targeted Therapy + Chemotherapy
  Interventions: Procedure: Interventional; Drug: Targeted Therapy (anti-VEGF); Drug: Immunotherapy + Targeted Therapy; Drug: Immunotherapy + Targeted Therapy + Chemotherapy; Other: This cycle is repeated every 21 days.

INTERVENTIONS:
Procedure: Interventional — Pancreatic tumor and liver metastases: TAC Liver metastases: For non-diffuse liver metastases with good blood supply: TACE
Drug: Targeted Therapy (anti-VEGF) — Apatinib 250 mg qd
Drug: Immunotherapy + Targeted Therapy — After 1-2 weeks Iparomlimab and Tuvonralimab (50 mg/2 mL) combined with Apatinib 250 mg qd
Drug: Immunotherapy + Targeted Therapy + Chemotherapy — After 3 weeks Iparomlimab and Tuvonralimab (50 mg/2 mL) on day 1 Albumin-bound paclitaxel 125 mg/m² on days 2 and 9 Gemcitabine 1000 mg/m² on days 2 and 9 Apatinib 250 mg qd
Other: This cycle is repeated every 21 days. — Interventional therapy is discontinued if imaging shows no enhancement of tumor vessels and is resumed only upon disease progression or until intolerable adverse reactions occur.

SUMMARY:
To evaluate the efficacy of arterial infusion chemotherapy and embolization combined with iparplidutol-volerilis (QL1706) as first-line treatment for pancreatic cancer liver metastases based on progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participate in this study, sign the informed consent form, demonstrate good compliance, and cooperate with follow-up visits.

  2. Male or female, aged 18 to 75 years. 3. ECOG performance status score of 0 to 1. 4. Expected survival ≥ 3 months. 5. Histologically or cytologically confirmed, previously untreated unresectable pancreatic ductal adenocarcinoma with liver metastases (TNM stage: IV).

  6. Must have measurable lesions according to RECIST 1.1 criteria. 7. No prior systemic therapy for pancreatic cancer or liver metastases, including chemotherapy, targeted therapy, or immunotherapy. (Note: Patients who received only one prior cycle of treatment, or oral targeted/chemotherapy agents for a cumulative duration ≤ 14 days, or those with recurrence more than six months after completing adjuvant chemotherapy may be considered for inclusion.) 8. Selective arterial catheterization and angiography demonstrate staining of pancreatic tumors and liver metastases. Patients with good tumor blood supply are eligible for this study.

  9. No local treatment (including transarterial chemoembolization/TACE, hepatic arterial infusion chemotherapy/HAIC, radiotherapy, radioembolization, or ablation, etc.) on target lesions within 28 days before the first dose of the study drug.

  10. Recovery from toxicities caused by prior therapies: ≥4 weeks since prior cytotoxic drugs, radiotherapy, or surgery, with wounds fully healed.

  11. No prior treatment with anti-PD-1, anti-PD-L1, anti-CTLA-4 antibodies, or CAR-T cell therapy.

  12. Adequate organ function must be confirmed within 28 days before the first dose (without transfusion or use of blood products, G-CSF, or other hematopoietic growth factors for correction within 14 days prior to laboratory tests):
  1. Absolute neutrophil count (ANC) ≥1.5×10⁹/L (without G-CSF support within 14 days).
  2. Platelets ≥100×10⁹/L (without transfusion within 14 days).
  3. Hemoglobin >9 g/dL (without transfusion or erythropoietin use within 14 days).
  4. Total bilirubin ≤1.5×ULN.
  5. AST and ALT ≤2.5×ULN.
  6. Serum creatinine ≤1.5×ULN and calculated creatinine clearance (Cockcroft-Gault formula) ≥60 mL/min.
  7. Adequate coagulation function, defined as INR or PT ≤1.5×ULN.
  8. Normal thyroid function, defined as TSH within normal range. If baseline TSH is abnormal, patients may still be enrolled if total T3 (or FT3) and FT4 are within normal limits.
  9. Cardiac enzymes within normal range (isolated laboratory abnormalities deemed clinically insignificant by the investigator are allowed).

  13. Males and females of childbearing potential must agree to use highly effective contraception from the time of signing the informed consent form until at least 5 months (for females) or 7 months (for males) after the last dose of the study drug. Women of childbearing potential must not be pregnant or breastfeeding.

Exclusion Criteria:

* **Subjects meeting any of the following criteria will be excluded from this study:**

  1. Diagnosis of another malignancy within 5 years prior to the first dose, unless cured (exceptions include radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ that has undergone radical resection).
  2. Currently participating in an interventional clinical study or having received other investigational drugs or devices within 4 weeks prior to the first dose.
  3. Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2 agents, or drugs targeting another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137).
  4. Poor tumor blood supply as observed during selective arterial catheterization and angiography of pancreatic tumors and liver metastases.
  5. Systemic treatment with Chinese herbal medicine with anti-tumor indications or immunomodulatory drugs within 2 weeks prior to the first dose.
  6. Active autoimmune disease requiring systemic treatment (e.g., disease-modifying agents, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency) is not considered systemic treatment.
  7. Current systemic corticosteroid therapy (excluding nasal sprays, inhalational, or other local corticosteroids) or any other form of immunosuppressive therapy within 7 days prior to the first dose.

     * Note:** Physiological doses of corticosteroids (e.g., ≤10 mg/day prednisone or equivalent) are permitted.
  8. Known history of allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
  9. Known hypersensitivity to iparomlimab and tuvonralimab or any excipients of the combined chemotherapy drugs used in this study.
  10. Insufficient recovery from toxicities and/or complications of prior interventions (i.e., not recovered to ≤ Grade 1 or baseline, excluding fatigue or alopecia) before starting treatment.
  11. Known history of human immunodeficiency virus (HIV) infection (i.e., positive for HIV 1/2 antibodies).
  12. Untreated active hepatitis B (defined as HBsAg positive with HBV-DNA copy number above the upper limit of normal [ULN] at the local laboratory).

      * Note:** Subjects with hepatitis B meeting the following criteria may be enrolled:

        1. HBV viral load < 1000 copies/mL (200 IU/mL) prior to the first dose. The subject must receive anti-HBV therapy throughout the study chemotherapy treatment period to prevent viral reactivation.
        2. Subjects who are anti-HBc (+), HBsAg (-), anti-HBs (-), and have undetectable HBV viral load do not require prophylactic anti-HBV therapy but require close monitoring for viral reactivation.
  13. Active HCV infection (HCV antibody positive with HCV-RNA levels above the lower limit of detection).
  14. Administration of a live vaccine within 30 days prior to the first dose (Cycle 1, Day 1).

      * Note:** Inactivated seasonal influenza vaccines administered by injection are permitted within 30 days prior to the first dose. However, live attenuated influenza vaccines administered intranasally are not permitted.
  15. Pregnant or breastfeeding women.
  16. Any severe or uncontrolled systemic disease, such as:

      1. Resting ECG showing significant and symptomatic abnormalities in rhythm, conduction, or morphology (e.g., complete left bundle branch block, second-degree or higher heart block, ventricular arrhythmia, or atrial fibrillation).
      2. Unstable angina, congestive heart failure, or chronic heart failure of New York Heart Association (NYHA) Class ≥2.
      3. Myocardial infarction within 6 months prior to enrollment.
      4. Poorly controlled hypertension (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg).
      5. History of non-infectious pneumonitis requiring corticosteroid treatment within 1 year prior to the first dose, or current clinically active interstitial lung disease.
      6. Active pulmonary tuberculosis.
      7. Active or uncontrolled infection requiring systemic therapy.
      8. Clinically active diverticulitis, abdominal abscess, or gastrointestinal obstruction.
      9. Liver diseases such as cirrhosis, decompensated liver disease, or acute or chronic active hepatitis.
      10. Poorly controlled diabetes (fasting blood glucose >10 mmol/L).
      11. Urinalysis showing protein ≥++ and confirmed 24-hour urine protein >1.0 g.
      12. Psychiatric disorders that may interfere with treatment compliance.
  17. Any medical history, condition, treatment, or laboratory abnormality that, in the investigator's judgment, may interfere with the trial results, prevent the subject from completing the study, or pose other potential risks making the subject unsuitable for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival（PFS） | Approximately 1 day after disease progression or death from any cause in cancer patients.
  The time from treatment initiation to disease progression or death from any cause in cancer patients.

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | Approximately 1 month after imaging examination
  The proportion of subjects who achieve complete response (CR) and partial response (PR) among the total subjects.
Disease Control Rate（DCR） | Approximately 1 month after imaging examination
  The proportion of patients with tumor shrinkage or stabilization maintained for a certain duration, including those with complete response (CR), partial response (PR), and stable disease (SD).
Duration of Response（DOR） | Approximately 1 day after the time from when the tumor first achieves an objective response (shrinkage or disappearance) to disease progression or death.
  The period from when a patient achieves an objective response (shrinkage or disappearance of the tumor) after treatment to disease progression or death.
Overall Survival (OS) | Approximately 2 years after last participant enrollment.
  The time from initial treatment to death from any cause
Adverse Event (AE) | Approximately 2 month after any treatment
  Type, incidence, grading (based on NCI-CTCAE v5.0 criteria), and duration of adverse event.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Maekawa A, Omiya K, Oba A, Inoue Y, Hirose Y, Kobayashi K, Ono Y, Sato T, Sasaki T, Ozaka M, Matsueda K, Mise Y, Takamatsu M, Shigematsu Y, Ito H, Saiura A, Sasahira N, Takahashi Y. Clinical implications of disappearing pancreatic cancer liver metastases: Lessons from colorectal liver metastases. Eur J Surg Oncol. 2025 May;51(5):109635. doi: 10.1016/j.ejso.2025.109635. Epub 2025 Jan 27. PMID 39879814